CLINICAL TRIAL: NCT05592067
Title: Effect of the Kinesiotaping on paın, Function and electrophysiologıcal Findings in Patient With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, medical doctor, asisst prof, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-16/146
Record Dates: First submitted 2022-10-14; First posted 2022-10-24 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: kinesiotaping; electrophysiological findings; carpal tunel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into 3 groups.Group A (kinesio taping with I tape technique + exercise to tendon and median nerve slipping), Group B (kinesio taping with button hole technique + exercise to tendon and median nerve slipping) and They will be divided into Group C (tendon and median nerve gliding exercise).
  In the first group, kinesio taping with the I tape technique described by Dr Kenzo Kase will be applied once a week, a total of 3 times, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  In the second group, kinesio taping with the Button hole technique defined by Dr Kenzo Kase will be applied once a week, 3 times in total, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  In the third group, exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor are blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- I tape technique (Active Comparator): I tape technique described by Dr Kenzo Kase will be applied once a week, a total of 3 times, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  Interventions: Other: I tape technique; Other: exercises
- Button hole technique (Active Comparator): Button hole technique defined by Dr Kenzo Kase will be applied once a week, 3 times in total, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  Interventions: Other: Button hole technique; Other: exercises
- exercises (Other): exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  Interventions: Other: exercises

INTERVENTIONS:
Other: I tape technique — I tape technique described by Dr Kenzo Kase will be applied once a week, a total of 3 times, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  Arms: I tape technique
Other: Button hole technique — Button hole technique defined by Dr Kenzo Kase will be applied once a week, 3 times in total, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.
  Arms: Button hole technique
Other: exercises — exercises will be taught to the patient and a total of 21 sessions will be applied once a day

SUMMARY:
The aim of this study is to compare the effectiveness of different kinesio taping techniques applied in carpal tunnel syndrome on pain, mobility, functional status and electrophysiological results and to investigate whether they are superior to the control group.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) was first described by Paget in 1854, and detailed information about its clinical course and surgical techniques were made by Phalen. Carpal tunnel syndrome (CTS) is a clinical picture consisting of symptoms resulting from compression of the median nerve in the carpal tunnel at the wrist level and is the most common entrapment neuropathy. Although it is due to idiopathic and secondary causes, the pathophysiology of CTS is not fully understood.

It is 3 times more common in women than in men. The fact that CTS occurs more frequently in the dominant hand supports the important role of hand activity in the emergence of the disease. Since the sensory branches of the median nerve innervate the first three fingers and half of the fourth finger, they typically complain of burning, pinprick, tingling and numbness in these fingers in CTS. In some cases, the pain may not match the normal sensory area of the median nerve in the hand.

The diagnosis of CTS is easily made by history and physical examination. Imaging and electrodiagnostic studies are helpful in confirming the diagnosis.

Treatment varies according to the degree of CTS. Different conservative treatment methods are used in the treatment of mild and moderate CTS. The most commonly used methods are splint, local corticosteroid injection (LCE), nonsteroidal anti-inflammatory drugs (NSAID) and conventional treatment agents (TENS, hotpack, ultrasound). Treatment modalities for edema and pain should not be ignored during the rehabilitation period. In this respect, kinesiotaping (KT) treatment, which is practical, comfortable and safe for the patient, is one of the complementary treatment modalities with positive clinical results.The purpose of the kinesiological taping (KB) method, developed by Kenzo Kase in the 1970s, is to support the muscle structures and increase their stability without limiting the range of motion of the joint. KB application is used with many indications such as pain, posture disorders, tendinitis bursitis, foot deformities, sports injuries, lymphedema and entrapment neuropathies.

Research on the use of kinesiotaping in the conservative treatment of carpal tunnel syndrome has increased in recent years. The data of our study will contribute to the literature in order to develop the right technique for kinesiotaping in the treatment of CTS.

The estimated number of volunteers expected to participate in the study was determined according to power analysis. The sample size of the study was determined by the GPower 3.1.9.6 program, and by using the finding in a similar study in the literature, it was used with 80% power and 5% margin of error to catch the medium effect size between dependent measurements. It was decided to work with a total of minimum 60 people, 20 in each group.Considering the patients who may be excluded from follow-up in the study, it is planned to start the study with 70 patients. The diagnosis of the disease will be made by clinical physical examination and enmg studies, and no additional technique will be required.

Patients will be randomly divided into 3 groups. (They will be selected by simple random sampling using the closed envelope method, and then Group A (kinesio taping with I tape technique + exercise to tendon and median nerve slipping), Group B (kinesio taping with button hole technique + exercise to tendon and median nerve slipping) and They will be divided into Group C (tendon and median nerve gliding exercise).

In the first group, kinesio taping with the I tape technique described by Dr Kenzo Kase will be applied once a week, a total of 3 times, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.

In the second group, kinesio taping with the Button hole technique defined by Dr Kenzo Kase will be applied once a week, 3 times in total, and the exercises will be taught to the patient and a total of 21 sessions will be applied once a day.

In the third group, exercises will be taught to the patient and a total of 21 sessions will be applied once a day.

Kinesiotaping application; It will be done by a physical therapist who has a kinesiology taping course certificate.

I tape technique: In this technique, an I tape is measured and cut from the heads of the metacarpals to the epicondyles of the humerus. The ends of the tape are cut and an x shape is obtained at the ends. The tape is folded to find the middle point, then the paper is torn and, starting from the middle point, the patient's wrist and elbow are moved to the extension of the palmaris longus entrance. distally, below the antecubital fossa, the lower forearm is adhered to the carpal tunnel region with mild-light (15-25%) tension. Taping is applied to the wrist from the dorsal side again with a field correction technique. With the wrist slightly flexed, the middle part of a 15-20 cm I tape is adhered to the distal radius and ulna from the dorsal face with very light-light (15-25%) tension. With one hand, the band is held over the styloid processes of the radius and ulna, and with the other hand, the wrist is extended. The remaining ends are cut and glued without tension, leaving a small gap between both ends.

Buttonhole: In this technique, a kinesio tape is measured and cut from the medial and lateral epicondyle level on the palmar side of the forearm, from the base of the proximal phalanges to the humerus epicondyles on the dorsal surface of the forearm. The tape is folded and the middle point is found there by making 2 short incisions and 2 holes through which it will pass between the 3rd and 4th fingers. (button holes) are obtained. The paper on the back of the tape is torn and the 2nd and 3rd fingers are passed through the holes. The patient's wrist is extended and radial deviation is brought, and the band is adhered to the medial epicondyle of the forearm with very light-mild (15-25%) tension. Then, the wrist is flexed and ulnar deviation is brought, and it is adhered to the lateral epicondyle with very light-mild (15-25%) tension. The last 3-5 centimeters are adhered without tension. Taping is applied to the wrist from the dorsal side again with a field correction technique. With the wrist slightly flexed, the middle part of a 15-20 cm I tape is adhered to the distal radius and ulna from the dorsal face with very light-light (15-25%) tension. With one hand, the band is held over the styloid processes of the radius and ulna, and with the other hand, the wrist is extended. The remaining ends are cut and glued without tension, with a small gap between both ends.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients aged 18-65 years who applied to Ahi Evran University Physical Medicine and Rehabilitation Outpatient Clinic and diagnosed with mild to moderate carpal tunnel syndrome by clinical and EMG
2. Patients who can correctly understand what is stated in the patient information form and have cooperation
3. Patients who consented to participate in the study according to the informed consent form

Exclusion Criteria:

1. Cervical radiculopathy
2. Polyneuropathy
3. Brachial plexopathy
4. Systemic corticosteroid use
5. History of fracture and trauma in the treated side forearm and wrist
6. Inflammatory rheumatic disease
7. Pregnant and lactating patients
8. Systemic diseases such as renal insufficiency, peptic ulcer, DM, hypothyroidism, coagulation disorder
9. Patients undergoing carpal tunnel syndrome surgery
10. Thoracic outlet syndrome
11. Thenar atrophy, severe carpal tunnel syndrome
12. The patient is reluctant or states that he cannot participate for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 0 (baseline)
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Visual Analog Scale | 3 th week
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Visual Analog Scale | 12 th week
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Hand grip strength | 0 (baseline)
  Jamar dynamometer will be used to measure hand grip strength. Jamar dynamometer measures static grip strength in pounds and kilograms. Measurements will be made with the patient in a sitting position, arm adducted, elbow flexed to 90 degrees, forearm in neutral position, as recommended by the American Association of Hand Therapists. Patients are asked to squeeze the dynamometer for at least 3 seconds with maximum contraction. 3 measurements are made with a 1 minute break between measurements. The average of 3 measurements is recorded in kilograms
hand grip strength | 3 th week
  Jamar dynamometer will be used to measure hand grip strength. Jamar dynamometer measures static grip strength in pounds and kilograms. Measurements will be made with the patient in a sitting position, arm adducted, elbow flexed to 90 degrees, forearm in neutral position, as recommended by the American Association of Hand Therapists. Patients are asked to squeeze the dynamometer for at least 3 seconds with maximum contraction. 3 measurements are made with a 1 minute break between measurements. The average of 3 measurements is recorded in kilograms
hand grip strength | 12 th week
  Jamar dynamometer will be used to measure hand grip strength. Jamar dynamometer measures static grip strength in pounds and kilograms. Measurements will be made with the patient in a sitting position, arm adducted, elbow flexed to 90 degrees, forearm in neutral position, as recommended by the American Association of Hand Therapists. Patients are asked to squeeze the dynamometer for at least 3 seconds with maximum contraction. 3 measurements are made with a 1 minute break between measurements. The average of 3 measurements is recorded in kilograms
electrophysiologıcal Findings | 0 (baseline)
  Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.
electrophysiologıcal Findings | 3 th week
  Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.
electrophysiologıcal Findings | 12 th week
  Median sensory nerve action potential amplitude, Compound muscle action potential amplitude, Median sensory distal latency, Median motor distal latency, Median sensory nerve conduction velocity, was evaluated by EMG.

SECONDARY OUTCOMES:
function | 0 (baseline)
  The Boston carpal tunnel questionnaire (BCTA) has been proposed for clinical standardization of CTS patients. It consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. A high mean score indicates that the patient's complaints are severe or that their functional capacity is insufficient. The symptom severity score is the average of the eleven questions and the functional capacity score of the eight questions.
function | 3 th week
  The Boston carpal tunnel questionnaire (BCTA) has been proposed for clinical standardization of CTS patients. It consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. A high mean score indicates that the patient's complaints are severe or that their functional capacity is insufficient. The symptom severity score is the average of the eleven questions and the functional capacity score of the eight questions.
function | 12 th week
  The Boston carpal tunnel questionnaire (BCTA) has been proposed for clinical standardization of CTS patients. It consists of nineteen questions and the answers are evaluated with a minimum of one and a maximum of five points. A high mean score indicates that the patient's complaints are severe or that their functional capacity is insufficient. The symptom severity score is the average of the eleven questions and the functional capacity score of the eight questions.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asisst Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kirşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geler Kulcu D, Bursali C, Aktas I, Bozkurt Alp S, Unlu Ozkan F, Akpinar P. Kinesiotaping as an alternative treatment method for carpal tunnel syndrome. Turk J Med Sci. 2016 Jun 23;46(4):1042-9. doi: 10.3906/sag-1503-4. PMID 27513402
- [Background] Yildirim P, Dilek B, Sahin E, Gulbahar S, Kizil R. Ultrasonographic and clinical evaluation of additional contribution of kinesiotaping to tendon and nerve gliding exercises in the treatment of carpal tunnel syndrome. Turk J Med Sci. 2018 Oct 31;48(5):925-932. doi: 10.3906/sag-1709-72. PMID 30384555
- [Result] Krause D, Roll SC, Javaherian-Dysinger H, Daher N. Comparative efficacy of the dorsal application of Kinesio tape and splinting for carpal tunnel syndrome: A randomized controlled trial. J Hand Ther. 2021 Jul-Sep;34(3):351-361. doi: 10.1016/j.jht.2020.03.010. Epub 2020 Sep 4. PMID 32893100
- [Derived] Sahin MA, Cigdem-Karacay B, Konar NM, Tuncay F. Comparison of the Effectiveness of 2 Different Kinesio Taping Techniques Added to Exercises in the Treatment of Carpal Tunnel Syndrome: Randomized Controlled Trial, Double-Blind, Parallel Groups. Arch Phys Med Rehabil. 2024 Sep;105(9):1657-1665. doi: 10.1016/j.apmr.2024.05.023. Epub 2024 Jun 6. PMID 38851555